CLINICAL TRIAL: NCT00079911
Title: An International, Randomized, Double-Blind, Placebo-Controlled Study of Valaciclovir for the Suppression and Episodic Treatment of Genital HSV Infection in HIV-Infected Persons With CD4+ Lymphocyte Count <100 Cells/mm3.
Brief Title: A Clinical Research Study For The Suppression And Treatment Of Genital Herpes Infection In HIV-Infected Persons
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Terminated
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 100181
Record Dates: First submitted 2004-03-18; First posted 2004-03-19 (Estimated); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Herpes Genitalis
Keywords: Herpes; Genital Herpes; HIV; HSV
MeSH Terms: conditions — Herpes Genitalis; Herpes Simplex | interventions — Valacyclovir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Suppressive + Episodic Therapy (Experimental): Valaciclovir (VAL) 500mg twice daily for 6 months, and episodic treatment with VAL 1000mg twice daily for 5 days or 10 days, when required for treatment of a genital herpes recurrence.
  Interventions: Drug: valacyclovir hydrochloride
- Episodic Therapy (Placebo Comparator): Matching placebo twice daily for 6 months, and episodic treatment with VAL 1000mg twice daily for 5 or 10 days, when required for treatment of a genital herpes recurrence.
  Interventions: Drug: valacyclovir hydrochloride

INTERVENTIONS:
Drug: valacyclovir hydrochloride — valacyclovir hydrochloride

SUMMARY:
This clinical research study will be an international trial evaluating the safety and effectiveness of a marketed drug compared to placebo (like a sugar pill) for the suppression of repeated genital herpes infections in HIV-infected subjects with CD4+ count <100 cells/mm3.

ELIGIBILITY:
Inclusion Criteria:

* CD4+ lymphocyte count <100cells/mm3 at the screening visit.
* Documented history of HIV infections
* Must have received stable, combination anti HIV drugs for at least 4 months immediately prior to participation, and per the investigator, are unlikely to require change in anti-HIV drugs during the six-month study.
* Laboratory confirmation of genital herpes (a positive Herpes Simplex Virus-2 antibody test).
* 3 or more outbreaks of genital herpes in the previous 12 months if not on genital herpes medicines currently.
* 3 or more outbreaks of genital herpes per year in the period prior to beginning of treatment for chronic genital herpes.

Exclusion Criteria:

* Kidney diseases.
* Liver diseases.
* Known allergic reactions to VALTREX (valaciclovir), ZOVIRAX (acyclovir), FAMVIR (famciclovir), or CYTOVENE (ganciclovir).
* Vomiting syndrome.
* Must be willing to discontinue taking current genital herpes medicines 1 week prior to participation.
* Active AIDS-indicator conditions, as defined by CDC Category C.
* Other protocol inclusion and exclusion criteria to be evaluated by the research physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2004-03-12 (Actual); Primary Completion 2004-10-15 (Actual); Study Completion 2004-10-15 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Up to 6 months
  The nature and incidence of adverse events, by treatment group, reported during the 6-month study will be summarized.

SECONDARY OUTCOMES:
Proportion of recurrence of genital HSV | Up to 6 months
  Secondary outcome measures are the proportion of subjects recurrence-free of genital HSV at 6 months, and the time to first culture-positive recurrence of genital HSV.
Time to first culture-positive recurrence of genital HSV | Up to 6 months
  Secondary outcome measures are the proportion of subjects recurrence-free of genital HSV at 6 months, and the time to first culture-positive recurrence of genital HSV.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- United States (3):
  - GSK Investigational Site, Altamonte Springs, Florida
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Boston, Massachusetts
- GSK Investigational Site, Darlinghurst, New South Wales, Australia
- GSK Investigational Site, Kowloon Bay, Hong Kong